CLINICAL TRIAL: NCT03747900
Title: Does Dry Needling Increase the Efficacy of Botulinum Toxin Injection in the Treatment of Poststroke Spasticity: A Randomized Controlled Study
Brief Title: Dry Needling and Botulinum Toxin in the Management of Poststroke Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MuratKOSEM
Record Dates: First submitted 2018-11-17; First posted 2018-11-20 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Spasticity, Muscle
Keywords: Needling, botulinum, toxin, spasticity, stroke
MeSH Terms: conditions — Muscle Spasticity; Stroke | interventions — Botulinum Toxins, Type A; Dry Needling

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BTX-A (Experimental): Patients underwent 200 U BTX-A injections in biceps brachii muscle.
  Interventions: Drug: Botulinum Toxin Type A
- BTX-A+Dry needling (Active Comparator): Dry needling was administered for 4 times in total after the BTX-A injection.
  Interventions: Combination Product: Botulinum Toxin Type A and dry needling.

INTERVENTIONS:
Drug: Botulinum Toxin Type A — 200 U Botulinum toxin type A injection in the spastic biceps brachii muscle.
  Arms: BTX-A
Combination Product: Botulinum Toxin Type A and dry needling. — Dry needling for 4 times in total in the spastic biceps brachii muscle after the Botulinum toxin type A injection.
  Arms: BTX-A+Dry needling

SUMMARY:
Stroke is a clinical picture that can result in loss of motor, sensory and cognitive functions or coma. Approximately 75% of stroke survivors develop disability and one of the causes of disability is the presence of spasticity. Effective treatment of spasticity accelerates functional recovery. Botulinum toxin type A (BTX-A) injection is a safe and effective method in the management of focal spasticity. As its effects over central and peripheral nervous system have been understood, dry needling has been recently introduced as the novel treatment of spasticity after stroke in clinical practice. Studies evaluating the efficacy of dry needling in the treatment of spasticity are limited in the literature and there is no data on the long-term efficacy of dry needling in current studies. On the other hand, the effects of dry needling when combined with other antispastic treatment modalities have not been investigated yet. In this study, the antispastic efficacy of dry needling applied with BTX-A injection was investigated.

DETAILED DESCRIPTION:
The study was designed as a prospective, randomized, single-blind study. Patients included in the study were selected from 59 stroke patients and randomized into two groups; BTX-A injections and exercise in BTX-A Group (n=15), and BTX-A injection and exercise, additionally with dry needling in BTX-A+Dry needling Group (n=15). All patients underwent 200 U BTX-A injections in biceps brachii muscle under sonographic guidance. Patients who were included in BTX-A+Dry needling Group underwent dry needling for 4 times in total following BTX-A injection, as the first one being administered immediately after the BTX-A injection, and the remaining three with a three-day interval (3rd, 6th and 9th days after BTX-A injection). Stretching exercises for the upper extremity spastic muscles and strengthening exercises for the antagonist muscles on the hemiplegic side were applied in both groups. Patients were followed for 3 months after injection. As a result, the data obtained in this study was compatible with the results that ultrasonography (US)-guided BTX-A injection to the upper extremity together with the rehabilitation program decreased the post-stroke spasticity, improved the upper extremity motor functions, and this improvement continued until 3 months after injection. In addition, dry needling combined with BTX-A injection and performed in a total of 4 sessions with three days intervals, contributes to the antispastic effect to start earlier, to be more effective and to maintain a longer-lasting effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first-time stroke
* To have Modified Ashworth Scale of 2 and 3 spasticity levels in the elbow flexor muscles of the hemiplegic side
* Not having any joint pathology that would prevent passive movements of the involved elbow joint

Exclusion Criteria:

* Having a mental problem
* Presence of cooperation-orientation limitation or neglect
* Use of an oral antispastic agent
* BTX-A application in the last 3 months
* Peripheral nerve injury in the affected side upper extremity
* Wound presence in the area where the procedure will be applied
* Patients with a contraindication for BTX-A application
* Patients with needle phobia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 6 months.
  The Modified Ashworth Scale (MAS) measures spasticity during passive soft-tissue stretching. MAS is a six-point ordinal scale for grading the resistance encountered during such passive muscle stretching. MAS grades spasticity as follows:
  0: No increase in muscle tone.
  1: Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is(are) moved in flexion or extension.
  1+: Slight increase in muscle tone, manifested by a catch followed by minimal resistance through the remainder of the range of motion but the affected part(s) is(are) easily moved.
  2: More marked increase in muscle tone through most of the range of movement, but the affected part(s) is easily moved.
  3: Considerable increases in muscle tone, passive movement difficult.
  4: Affected part(s) is (are) rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)